CLINICAL TRIAL: NCT05129813
Title: Improving Treatment and Recovery Services for Individuals With Opioid Problems and Their Family Members
Brief Title: Improving Treatment and Recovery Services for Individuals With Opioid Problems
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Howard University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Boston University (Other); University of Maryland, College Park (Other); Yale University (Other); Unity Health Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-18-MED-38; 3UG1DA013034-20 (NIH)
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Counseling
Keywords: Opioid Use Disorder; Behavioral Counseling; Peer Recovery Specialist; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Buprenorphine MOUD in FQHC: Participants receiving buprenorphine treatment and Recovery Guide counseling in a Federally Qualified Health Center. Recovery Guide counseling is provided weekly.
  Interventions: Behavioral: Recovery Guide Counseling
- Telemedicine Provision of Buprenorphine MOUD in a community site: Participants receiving buprenorphine treatment provided by telemedicine from a hub clinic and Recovery Guide counseling in a church or faith-based community organization. Recovery Guide counseling is provided weekly.
  Interventions: Behavioral: Recovery Guide Counseling

INTERVENTIONS:
Behavioral: Recovery Guide Counseling — Recovery Guide Counseling is a 12-session psychoeducational and behavioral counseling intended for delivery by Peer Recovery Specialists, community health workers, or other personnel without advanced training in counseling

SUMMARY:
Participants include persons receiving buprenorphine treatment and Recovery Guide counseling in a Federally Qualified Health Center or buprenorphine treatment by telemedicine and Recovery Guide counseling in a church or faith-based community organization. Participants are interviewed at the outset of treatment, after 4 to 6 weeks, and then at 10 to 12 weeks of treatment. The study is an observational study aimed at evaluating the experiences and response to treatment of participants.

DETAILED DESCRIPTION:
Participants include persons receiving buprenorphine treatment and Recovery Guide counseling in a Federally Qualified Health Center or buprenorphine treatment by telemedicine and Recovery Guide counseling in a church or faith-based community organization. Participants are interviewed at the outset of treatment, after 4 to 6 weeks, and then at 10 to 12 weeks of treatment. The study is an observational study aimed at evaluating the experiences and response to treatment of participants. Interviews use a semi-structured format assessing current and past opioid and other substance use, adherence to buprenorphine, and experiences with the counseling and other services provided.

ELIGIBILITY:
Inclusion Criteria:

* Opioid use disorder
* Initiating buprenorphine treatment

Exclusion Criteria:

* Inability to understand the study protocol or assessment questions
* Severe medical or psychiatric co-morbidity, including active psychosis, high risk for suicide, or medical contraindications to buprenorphine (e.g., allergy or sensitivity to buprenorphine),
* Currently (or in the past 30 days) receiving MAT for OUD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential participants will be recruited through posters, flyers, or word-of-mouth or information provided to them by neighborhood or community agencies or organizations or referred by their medical provider.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Retention | 12 weeks
  Proportion of participants continuing to receive buprenorphine treatment at 12 weeks

SECONDARY OUTCOMES:
Medication adherence | 12 weeks
  Percent days self-reported medication adherence
Treatment satisfaction | 12 weeks
  Self-reported satisfaction with treatment

OTHER OUTCOMES:
Self-reported opioid and other drug use | 12 weeks
  Self-reported drug use
Health-related quality of life | 12 weeks
  Self-reported health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schottenfeld, M.D., Principal Investigator — Howard University
Locations (1):
- Howard University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No